CLINICAL TRIAL: NCT05884515
Title: Community Study to Evaluate the Performance of COVID-19 Frequent Antigen Testing at Home Through Digital Health Reporting
Brief Title: Evaluation of Home Use COVID-19 Frequent Antigen Testing and Data Reporting
Acronym: Chelsea_MA
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: IDX20 Inc (Industry)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: COVID-19 frequent testing; 4U24MD016258-02 (NIH)
Record Dates: First submitted 2023-05-30; First posted 2023-06-01 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: COVID-19 Respiratory Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- PCR comparator (Other): Another molecular test like PCR will be done to confirm the positive and negative antigen test
  Interventions: Diagnostic Test: SARS CoV-2 antigen tests

INTERVENTIONS:
Diagnostic Test: SARS CoV-2 antigen tests — The intervention is to compare antigen tests

SUMMARY:
The current standard of care for diagnostic of SARS-CoV-2 infection involves sample collection which is then prepared and measured via real time-polymerase chain reaction (RT-PCR). This process is time consuming and dependent on expensive instrumentation and trained technicians to perform both the sample preparation and assay. In many cases, sample turn-around times can take hours to several days. There are no established monitoring nationwide protocols for COVID-19 prevention of infection. Due to the lack of such protocols, this study will provide the proper experience to design a safe monitoring schema of asymptomatic cases of COVID-19.

Self-testing using currently available RDT has a high specificity and relatively high sensitivity to identify individuals with a high probability of contagiousness. Therefore, we intend to use these RDT (Rapid diagnostic tests) for other use.

There are several studies that point to the importance of the use of RDTs to monitor COVID-19 (3). The recent metadata indicate that the performance of the antigen test is crucial for obtaining good results to detect positive cases. We have already validated in the laboratory and using relevant clinical samples several different labels of antigen tests and we have compared them with already approved USA FDA antigen tests to confirm their performance prior to using them in this study.

This project aims to monitor once a week the presence of SARS CoV-2 antigens using anterior nares (AN) swab self-process, executing the test and recording of the result, immediately after.

The lack of affordable diagnostic tests which can detect the presence of SARS-CoV-2 in the general population which can give near real-time results is one critical missing control intervention in USA for the control of the pandemic and the spread of this disease. As public health restrictions begin to ease and people return to normal activities, while the COVID-19 pandemic is still a threat, a rapid diagnostic assay that does not require the sophisticated laboratory equipment and techniques could provide a significant advantage to screen asymptomatic individuals. The routine use of such rapid tests is a key element to show efficacy of protocol. We adjusted to once a week testing based on the medium to low risk of the elderly population of this study.

The list of rapid nucleoprotein tests utilized in the current study are: NETO Corona test, Novir INSTA-TM COVID-19 Rapid Antigen test, COVICHEK COVID-19 Ag Test, SpectraBiotech COVID-19 track antigen test, Blandford Biotech AS-15™ Rapid Antigen Detection Kit SARS-CoV-2 Test (Colloidal Gold Method), Abbott BinaxNow tests.

BACKGROUND

The SARS-CoV-2 Direct Antigen Rapid Test ("Lateral flow") is an immunoassay developed for the qualitative detection of SARS-CoV-2 viral particles/secreted protein in anterior nasal swabs and/or saliva samples from both asymptomatic and suspected participants with COVID-19 infection. Lateral flow strips are printed with a monoclonal antibody that binds the signature SARS-CoV-2 viral particles/protein (Test line) and a control antibody (Control line) for quality control. A second monoclonal antibody is attached to gold nanoparticles (conjugate) and quencher buffer, and mixed with the nasal sample. The SARS-CoV-2 nucleocapsid protein attach to both antibodies resulting in a visual line on the test strip within 15 minutes. Prior experience in the detection of virus and viral proteins via antibody binding using lateral flow have been done through IDx20, Inc. The Housing Authority and the Public Health Department of the City of Chelsea will be overseeing this study.

DETAILED DESCRIPTION:
The protocol will be deployed at three sites in the same geographical location. The design encompasses weekly monitoring of asymptomatic, non- disease populations, confirmed by RT-PCR for presumed positive cases. Each positive case will be followed with daily antigen testing and matched RT-PCR testing for 8 consecutive days in accordance with the CDC's stay-at-home protocol, the positive case will quarantine according to public policy. In addition to asymptomatic participants, participants presenting with a positive The antigen tests that will be utilized are all commercial final products with a CE mark.

All antigen tests utilized are close to identical procedure. Appendix 1 shows the instructions for use of each of the tests. All tests determined nucleoprotein of SARS CoV-2 in a qualitative manner.

Participants are not expected to participate beyond sample collection and processing of rapid antigen test as part of the study. The collection of one anterior nares sample is done once a week. A second nasal swab will be done once a sample indicates presumptive positive for COVID-19. At the end of 4 months of the study we will provide a rate of positive cases over time, and a positive agreement value over 8 days of testing of a positive case. The data will include a Positive Percent Value (PPV) and potentially expand to provide a NPV when negative samples are sent to the CLIA lab to determine the specificity of the tests.

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Individuals 12 year of age or older
2. Provision of paper-consent form and acceptance of participating on a volunteer basis.

Eligible affiliates are individuals who are associated to the member communities of each site and who are identified and consented into the study. These may be individuals who are in close contact with the member community and thus seen as peripheral community members.

* Subjects will be approached by research staff to determine if they would be interested in participating in this study. If willing, a qualified study team member will consent the subject. The electronic system will keep the information about approval of the informed consent by participant. We will also keep a record of the paper and a digital photo of the same document.
* Study staff will provide instructions to participants in the sample collection procedures on site to ensure proper self-sample collection and to minimize the risk of sample contamination. At the time of initial training. The participant will be using a self-swabbing process to obtain the NA sample. If we encounter an impediment for self-swabbing, the process will be done by assisting the participant.
* There will be 3 sites in the same geographical location. The design encompasses weekly monitoring of asymptomatic, non- disease populations by antigen test.The positive case will be followed with daily PCR / antigen test testing for 8 consecutive days in accordance with the CDC's stay-at-home protocol, each quarantine period will be completed. This screening will be used for assessing positive cases and confirming using a CLIA lab authorized molecular test.
* All materials part of the COVID-19 antigen test kit will be provided by the sponsor (Manufacturers provide the test to the sponsors). The test cassettes will be kept at Room Temperature.

SCIENTIFIC RATIONALE FOR STUDY DESIGN

The testing of asymptomatic cases to mitigate COVID-19 Pandemic requires frequent use in the population. Lateral flow bioassays are relatively inexpensive to manufacture, easy to store, and easy for front line use in public setting.

END OF STUDY DEFINITION

Participants are not expected to participate beyond frequent sample collection and processing of rapid antigen test as part of the study. The collection of anterior nares sample will be done once a week, as well as daily testing for up to 8 days in case of positive PCR result.

STUDY POPULATION

INCLUSION CRITERIA

1. Individuals age 12 or older
2. Provision paper-consent and acceptance of participating on a volunteer basis.

Up to 450 residents at:

Margolis Apartments (Federal Elderly/Disabled) - A 152- unit thirteen-story brick structure for elderly and/or disabled residents

Buckley Apartments (State Elderly/Disabled) - Located at 14 Bloomingdale Street has 210 one-bedroom apartments

Housing at 242 Walnut Street (State Elderly/Disable 40 Units

Affiliates are individuals who are associated to the member communities of The Chelsea Project sites and who are identified and consented into the study. These may be individuals who are in close contact with the member community and thus seen as peripheral community members.

EXCLUSION CRITERIA

If the participant requires medical urgent attention at the site of collection.

PARTICIPANT DISCONTINUATION/WITHDRAWAL

DISCONTINUATION OF STUDY SAMPLE EVALUATION

Subjects may withdraw at any time and request that their samples not be processed.

STUDY ASSESSMENTS AND PROCEDURES

STUDY PROCEDURES

All materials will be provided by the sponsor (IDx20-CCI) along with the co-sponsors owners of the test cassettes. The test cassettes should be kept at Room Temperature until use and in an indoor environment.

1. Subjects will be approached by research staff to determine if they would be interested in participating in this study. If willing, a qualified study team member will conduct a paper or e-informed consent process with the subject. The detailed procedure to conduct the test will be provided (insert) for each type of test each week. In two lenguages. The electronic system will populate the information about approval of the verbal informed consent by participant and it will provide a digital step by step instructions.
2. Study staff will provide support to participants to obtain the instructions and materials for sample collection procedures on site at each of the Chelsea Project sites to ensure proper sample collection and to minimize the risk of sample contamination.
3. The building administrator will have information of a presumptive positive case. Each site will follow their approved procedures for quarantine once the participant has been confirmed by RT-PCR. The participant will be tested at home each day after contracting COVID-19 for the following 8 days. The samples for PCR confirmation will be collected at home and sent to a CLIA lab.

Participant confidentiality and privacy is strictly held in trust by the participating investigators, their staff, and the sponsor(s) and their interventions. This confidentiality is extended to cover testing of biological samples in addition to any clinical information relating to participants. Therefore, the study protocol, documentation, data, and all other information generated will be held in strict confidence. No information concerning the study, or the data will be released to any unauthorized third party without prior written approval of the sponsor.

The study monitor, other authorized representatives of the sponsor, representatives of the Institutional Review Board (IRB), regulatory agencies or pharmaceutical company supplying study product may inspect all documents and records required to be maintained by the investigator, including but not limited to, medical records (office, laboratory facility).

The study participant's contact information will be securely stored at each site for internal use during the study. At the end of the study, all records will continue to be kept in a secure location for as long a period as dictated by the reviewing IRB, Institutional policies, or sponsor requirements.

Study participant research data, which is for purposes of statistical analysis and scientific reporting, will be transmitted to and stored at the The Chelsea Project server. A designed application will be used for the collection of cassette result images. This will not include the participant's contact or identifying information and includes participant ID numbers only. Rather, individual participants and their research data will be identified by a unique study identification number. The study data entry and study management systems used by study sites and by sponsor research staff will be secured and password protected. At the end of the study, all study databases will be de-identified and archived at the sponsor facilities.

FUTURE USE OF STORED SPECIMENS AND DATA

The nasal swab collected in saline will be required for RT-PCR confirmation, these samples will be stored at the CLIA lab (EcoLaboratory. Acton Ma). After the study is completed, the de-identified, archived data will be for use by other researchers as determined by sponsor only.

The data of the study could be used for research purposes.

During the conduct of the study, an individual participant can choose to withdraw consent to have biological specimens stored for future research. However, withdrawal of consent with regard to bio sample storage may not be possible after the study is completed.

ELIGIBILITY:
Inclusion Criteria:

* older than 12 years of age

Exclusion Criteria:

* critical ill

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2021-12-13 (Actual); Primary Completion 2023-11-21 (Estimated); Study Completion 2023-11-21 (Estimated)

PRIMARY OUTCOMES:
Diagnostic tests results positive or negative | 12 months
  PPA and NPA are calculated when comparing antigen tests to PCR results

CONTACTS AND LOCATIONS:
Overall Officials: Irene Bosch, PhD, Principal Investigator — IDX20 Inc
Locations (1):
- Chelsea Housing Authority, Chelsea, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
We will establish secure data transfer for all fields and data collected

REFERENCES:
- [Background] Harmon A, Chang C, Salcedo N, Sena B, Herrera BB, Bosch I, Holberger LE. Validation of an At-Home Direct Antigen Rapid Test for COVID-19. JAMA Netw Open. 2021 Aug 2;4(8):e2126931. doi: 10.1001/jamanetworkopen.2021.26931. PMID 34448871
- [Background] Kirby JE, Riedel S, Dutta S, Arnaout R, Cheng A, Ditelberg S, Hamel DJ, Chang CA, Kanki PJ. Sars-Cov-2 antigen tests predict infectivity based on viral culture: comparison of antigen, PCR viral load, and viral culture testing on a large sample cohort. Clin Microbiol Infect. 2023 Jan;29(1):94-100. doi: 10.1016/j.cmi.2022.07.010. Epub 2022 Jul 19. PMID 35863629
- See also: Website of Sponsor — https://www.idx20.us